

FARAPULSE\_PersAFOne II SAP V1.0

**Sponsor:** FARAPULSE

Device: FARAPULSE CARDIAC

ABLATION SYSTEM

PLUS

**Protocol Nr: CS1335** 

**REVISION B** 

ICON Project Nr:5326/0019

# Feasibility Study of the FARAPULSE Cardiac Ablation System Plus in the Treatment of Persistent Atrial Fibrillation PersAFOne II

Statistical Analysis Plan

| Versions | Date | Documents used | Statistical Lead | Senior Reviewer |
|---|---|---|---|---|
| V1.0 | 24/03/2023 | - CS1335_Rev A to Rev B<br>PersAFOne II Clinical<br>Protocol_19May2022.pdf | Najeh DAABEK | Marie Christine<br>REYMOND |
| | | - PersAFOnell_Annotated<br>CRF_revC_21Sep2022.<br>pdf | | |
| | | - PersAFOnell_Annotated<br>CRF_CEC.pdf | | |
| | | - Jan 2022_Endpoints for<br>Persafone CZ II.xlsx | | |
| V0.3 | 17/03/2023 | - CS1335_Rev A to Rev B<br>PersAFOne II Clinical<br>Protocol_19May2022.pdf | Najeh DAABEK | Marie Christine<br>REYMOND |
| | | - PersAFOnell_Annotated<br>CRF_revC_21Sep2022.<br>pdf | | |
| | | - PersAFOnell_Annotated<br>CRF_CEC.pdf | | |
| | | - Jan 2022_Endpoints for<br>Persafone CZ II.xlsx | | |

Sponsor:
BOSTON SCIENTIFIC, INC.
Way Marlborough
MA 01752
USA
France

CRO: ICON Clinical Research SARL Immeuble Le Capitole 55 Avenue des Champs Pierreux 92000 Nanterre



FARAPULSE\_PersAFOne II SAP V1.0

Sponsor: FARAPULSE

Device: FARAPULSE CARDIAC

ABLATION SYSTEM

PLUS

Protocol Nr: CS1335

REVISION B

ICON Project Nr:5326/0019

| V0.2 | 09/03/2023 | - | CS1335_Rev A to Rev B<br>PersAFOne II Clinical<br>Protocol_19May2022.pdf | Najeh DAABEK | Marie<br>REYMOND | Christine |
|---|---|---|---|---|---|---|
| | | - | PersAFOnell_Annotated CRF_revC_21Sep2022. pdf | | | |
| | | - | PersAFOnell_Annotated CRF_CEC.pdf | | | |
| | | - | Jan 2022_Endpoints for<br>Persafone CZ II.xlsx | | | |
| V0.1 | 06/03/2023 | • | CS1335_Rev A to Rev B<br>PersAFOne II Clinical<br>Protocol_19May2022.pdf | Najeh DAABEK | Marie<br>REYMOND | Christine |
| | | - | PersAFOnell_Annotated CRF_revC_21Sep2022. pdf | | | |
| | | - | PersAFOnell_Annotated CRF_CEC.pdf | | | |
| | | - | Jan 2022_Endpoints for<br>Persafone CZ II.xlsx | | | |

Sponsor: BOSTON SCIENTIFIC, INC. Way Marlborough MA 01752 USA France CRO: ICON Clinical Research SARL Immeuble Le Capitole 55 Avenue des Champs Pierreux 92000 Nanterre



FARAPULSE\_PersAFOne II SAP V1.0

**Sponsor:** FARAPULSE

Device: FARAPULSE CARDIAC

ABLATION SYSTEM

PLUS

Protocol Nr: CS1335

**REVISION B** 

ICON Project Nr:5326/0019

# SIGNATURE PAGE

# PERSAFONE II V1.0

# FARAPULSE, INC

| Name | Position | Date | Signature |
|---|---|---|---|
| Anitha Achyutha | Director, Clinical | | itha Achyutha<br>Mar 2023 15:50:02 UTC (Z)<br>t |
| Annelies Vanderper | EU Senior Manager<br>Clinical Trials | Annelie Vanderper REASON: I approve this docum | Annelies Vanderper<br>24 Mar 2023 10:08:19 UTC)(2<br>nt |

# **ICON CLINICAL RESEARCH SARL**

| Name | Position | Date | Signature |
|---|---|---|---|
| Marie-Christine<br>REYMOND | Senior Manager,<br>Biostatistics | Marie Christine Reymond 27 r | |
| Najeh DAABEK | Biostatistician II | 8116ca69-9263-4d28-b2da-9a8a4546320 Najeh Daabek 24 | jeh Daabek<br>Mar 2023 09:25:38 UTC (Z) |

REASON: I approve this document d0fe0951-4e46-41f5-9c58-01c89f6dec07



FARAPULSE\_PersAFOne II SAP V1.0 PERSAFONE II V1.0


# **TABLE OF CONTENTS**

| Lis | t of ab | breviati | ons and definition of terms | 5 |
|---|---|---|---|---|
| 1. | Over | view | | 6 |
| | 1.1. | Study C | bjective | 6 |
| | 1.2. | • | esign | |
| | 1.3. | - | lan | |
| | 1.5. | 1.3.1. | Sample Size | |
| | | 1.3.2. | Patient's Follow-up. | |
| | | 1.3.3. | Study Device use | |
| | | 1.3.4. | Study Assessments | |
| 2. | Statis | stical m | ethods | 7 |
| | 2.1. | | Statistical Considerations | |
| | 2.1. | 2.1.1. | Time Points Definition | |
| | | 2.1.2. | Handling Missing Data | |
| | | 2.1.3. | Descriptive Statistics in Summary Tables | |
| | | 2.1.4. | Inferential Analysis | |
| | | 2.1.5. | Data Listings | 8 |
| | 2.2. | Sample | size calculation. | 8 |
| | 2.3. | | s Sets | |
| | 2.3. | 2.3.1. | Definition of patient populations | |
| | | 2.3.2. | Protocol Deviations | |
| | | 2.3.1. | Databases | |
| | 2.4. | Statistic | al Analyses | 10 |
| | | 2.4.1. | Patient Disposition and Follow-up | |
| | | 2.4.2. | Baseline Patient Characteristics. | |
| | | 2.4.3. | Index Procedure | 10 |
| | | 2.4.4. | Follow-up at remapping procedure | 11 |
| | | 2.4.5. | 6 and 12 Months follow up | |
| | | 2.4.6. | Feasibility Analysis | |
| | | 2.4.7. | Additional endpoints | |
| | | 2.4.8. | Safety Endpoint | |
| | | 2.4.9. | Concomitant Medications | |
| | 2.5. | Derived | Criteria Calculation | 13 |
| 3. | Statis | stical So | ftware | 25 |
| 4. | Statis | stical tal | oles, Listings and Graphs (Table of contents) | 25 |
| | 4.1. | | al Tables | |
| | | 4.1.1. | Table 1. Subject enrollment per Site | |
| | | 4.1.2. | Table 2. Demographics | |
| | | 4.1.3. | Table 3. Baseline Medical History | 26 |
| | | 4.1.4. | Table 4. Procedure | |
| | | 4.1.5. | Table 5. Remap at 60 Days | |
| | | 4.1.6. | Table 6. Per Remapped Veins Analysis | |
| | | 4.1.7. | Table 7. Arrythmia Recurrence at 12 Months | |
| | | 4.1.8. | Table 8. Primary Safety Endpoint –Composite Safety Endpoint (CSE) | |
| | | 4.1.9. | Table 9. Primary Feasibility Endpoint – Acute Procedural Success (ITT population) | |
| | | 4.1.10.<br>4.1.11. | Table 10. Primary Feasibility Endpoint – Acute Procedural Success (PP population) Table 11. Additional Endpoints | |
| | | 4.1.11. | Table 11. Additional Endpoints | |
| | | T.1.1∠. | 14010 12. Decondary Darety Emaponium | |



FARAPULSE\_PersAFOne II SAP

PERSAFONE II

V1.0


| | 4.1.13. | Table 13. Secondary Feasibility Endpoints | |
|---|---|---|---|
| | 4.1.14. | Table 14. Adverse Events (AEs) (not including SAEs) | |
| | | Table 15. Serious Adverse Events (SAEs) | |
| | | Table 16. All Deaths | |
| | | Table 17. Protocol Deviations according investigator without COVID-19 | |
| | | Table 18. Protocol Deviations according investigator with COVID-19 | |
| | 4.1.19. | Table 19. Device Deficiency Summary Table | 38 |
| 4.2. | Listings | | 39 |
| | 4.2.1. | Listing 1: Patients populations, reasons of non-inclusion in the different population, | |
| | | withdrawals and follow-up duration | |
| | 4.2.2. | Listing 2: Protocol deviations according the investigator | 39 |
| | 4.2.3. | Listing 3: Demographics at baseline | 39 |
| | 4.2.4. | Listing 4: AF History | 39 |
| | 4.2.5. | Listing 5: Medical History (1/3) | 39 |
| | 4.2.6. | Listing 6: Medical History (2/3) | |
| | 4.2.7. | Listing 7: Medical History (3/3) | 39 |
| | 4.2.8. | Listing 8: Procedure data (1/4) | 39 |
| | 4.2.9. | Listing 9: Procedure data (2/4) | 39 |
| | 4.2.10. | Listing 10: Procedure data (3/4) | 39 |
| | 4.2.11. | Listing 11: Procedure data (4/4) | 39 |
| | 4.2.12. | Listing 12: Additional Ablation | 39 |
| | 4.2.13. | Listing 13: Chronic Procedural Success at remap | 39 |
| | 4.2.14. | Listing 14: Primary Safety endpoints | 39 |
| | | Listing 15: Device Deficiencies | |
| | 4.2.16. | Listing 16: Adverse events according CEC review | 39 |
| | | Listing 17: Serious adverse events according CEC review | |
| | 4.2.18. | Listing 18: Concomitant Medications | 39 |
| 4.3. | Graphs. | | 40 |
| | 4.3.1. | Graph 1: Patient disposition | |
| | 4.3.2. | Graph 2: Freedom from AF/AFL/AT on ADDs | |
| | 4.3.3. | Graph 3: Freedom from AF/AFL/AT off ADDs | |
| | 4.3.4. | Graph 4: Freedom from AF on AADs | |
| | 4.3.5. | Graph 5: Freedom from AF off AADs | |
| | 4.3.6. | Graph 6: Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days | |
| | 4.3.7. | Graph 7: Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days o AADS | |
| | 4.3.8. | Graph 8: Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days o AADS | ff |
| | 4.3.9. | Graph 9: Freedom from AF, no DCCV>90 days, no RF, no ablation >90 days on AADs | |
| | 4.3.10. | Graph 10: Freedom from AF, no DCCV>90 days, no RF, no ablation >90 days off AADs | |
| | 4.3.11. | Graph 11: Death | |



FARAPULSE\_PersAFOne II SAP V1.0 PERSAFONE II V1.0 Page 6 /42

## LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

| AAD | Antiarrhythmic drug |
|--------|--------------------------------|
| ABL | Ablation |
| AE | Adverse event |
| AF | Atrial fibrillation |
| AFL | Atrial Flutter |
| BMI | Body mass index |
| CPS | Chronic Procedural Success |
| СТ | Computed tomography |
| CSE | Composite Safety Endpoint |
| СТІ | Cavotricuspid isthmus |
| DCCV | Direct current cardioversion |
| ІПТ | Intention to treat |
| LA | Left atrium or left atrial |
| MRI | Magnetic resonance imaging |
| SAP | Statistical analysis plan |
| PEF | Pulsed electric field |
| PersAF | Persistent atrial fibrillation |
| PP | Per protocol |
| PT | Preferred term |
| PV | Pulmonary vein |
| SAE | Serious adverse event |
| SOC | System Organ system |
| TIA | Transient ischemic attack |



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


## 1. OVERVIEW

This statistical analysis plan (SAP) describes the planned statistical analyses of the data collected during the clinical study PersAFOne II.

This SAP provides additional details concerning the statistical analyses outlined in the protocol (CS1335\_Rev A to Rev B PersAFOne II Clinical Protocol\_19May2022).

## 1.1. Study Objective

The objective of this safety and feasibility study is to assess whether the endocardial creation of electrically nonconductive lesions via PEF catheter ablation applied using the FARAPULSE Cardiac Ablation System Plus is a feasible and safe treatment for Persistent atrial fibrillation (PersAF) and associated Atrial flutter (AFL)

## 1.2. Study Design

This is a prospective, multi-center, unblinded single arm safety and feasibility study. Subjects will undergo percutaneous PEF ablation for pulmonary vein isolation and at the clinical discretion of the investigator receive PEF (Pulsed electric field) ablation of additional arrhythmogenic locations. Subjects will be followed at 30 days, 60 days, 6 months and 12 months for adverse events, recurrence of arrhythmia after a 90-day Blanking Period and other relevant outcome measures.

#### 1.3. Study Plan

### 1.3.1. Sample Size

Up to 60 subjects in total will be enrolled at up to four sites in this clinical safety and feasibility study. Approved sites will enroll at least 5 and not more than 30 subjects.

#### 1.3.2. Patient's Follow-up

7 visits are scheduled:

- Visit 1: Baseline
- Visit 2: Index Procedure
- Visit 3: Pre-Discharge
- Visit 4: 30-Day Visit
- Visit 5: 60-DayVisit and Remapping Procedure
- Visit 6: 6-MonthVisit
- Visit 7: 12-MonthVisit

### 1.3.3. Study Device use

The FARAPULSE Cardiac Ablation System Plus is indicated for the treatment of drug refractory, recurrent, symptomatic persistent atrial fibrillation.

The FARAPOINT Pulsed Field Ablation Catheter is used as an adjunctive device in the endocardial treatment of persistent atrial fibrillation with the following intended uses:

• Gap ablation to complete electrical isolation of the pulmonary veins,



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


- · Focal ablation of cardiac arrhythmias, and
- Creation of ablation line between the inferior vena cava and the tricuspid valve.

## 1.3.4. Study Assessments

The following flowchart applies to the study:

| Assessment | Baseline | Procedure | Pre-Discharge | 30-Days Post-<br>Procedure (± 7<br>days) | 60-Days (± 15 days) | 6-Month<br>(180 ± 30<br>days) | 12-Month<br>(365 ± 30<br>days) | Unscheduled |
|---|---|---|---|---|---|---|---|---|
| Medical History, CHA2DS2-VASc | X | | | | | | | |
| AFD and Anticoagulant Medications | X | | X | Х | x | Х | X | Х |
| Symptoms of recurrent arrhythmia | | | | Х | x | Х | X | Х |
| History of cardioversions, ablations,<br>hospital admissions since last visit | | | X | Х | x | х | X | Х |
| Pregnancy test (for females of<br>childbearing potential) | X | x | | | /x | X <sup>4</sup> | X <sup>4</sup> | |
| 12-lead ECG | X | | X | X | x | X | X | X |
| 24-Hour Continuous ECG Monitor<br>(e.g., Holter) | | | | | / | х | X | |
| Cardiac CT/MRI for LA and PV dimensions | X | | | | Х | | | |
| Mediastinal MRI | | | $\mathbf{X}^{1}$ | | | | | |
| TEE or other imaging modality (to exclude left atrial thrombus) | X | | | | | | | |
| Electroanatomical Mapping | | X | / | | X | | | |
| Event Monitor readiness/compliance | | | | | X | X | X | X |
| NIHSS | X | | / X | | | | | |
| Neurologic exam | | | X2 | | | | | |
| NYHA Classification | X | , | X | X | X | X | X | X |
| Fluoroscopic Examination of<br>Diaphragm | | x | | | X if remapped,<br>X <sup>3</sup> if not | $X^3$ | X <sup>3</sup> | |
| Adverse Events | , | X | X | X | X | X | X | X |

## 2. STATISTICAL METHODS

#### 2.1. General Statistical Considerations

#### 2.1.1. Time Points Definition

Baseline data is defined as the last available observation recorded before the first study device exposition for the patient.

Visit(n) data is defined as the last available observation on or before the Visit(n) time point following the first study device exposition for the patient.

## 2.1.2. Handling Missing Data

In order to provide unbiased and informative findings, no replacement of missing values is planned for any parameters. Analyses is performed with all available data only.

Data collected by the Investigators and reviewed by the Clinical Event Committee (CEC):

When the data are collected by the investigators and reviewed by the CEC, the analysis will be as follows:

 The data reviewed by the CEC will prevail and will be analyzed with no replacement of missing data from the CEC with the data collected by the investigator



FARAPULSE\_PersAFOne II SAP V1.0 PERSAFONE II V1.0


## 2.1.3. Descriptive Statistics in Summary Tables

- Continuous variables will be summarized using standard quantitative statistics: number of nonmissing observations, mean, standard deviation, median, quartiles and range (minimum and maximum observed values). The number of missing observations will also be specified.
- Categorical variables will be summarized using classical frequency statistics: number of nonmissing observations and percentages by categories. Percentages will be calculated on the number of non-missing observations and will be displayed using one decimal. The number of missing observations will also be specified

## 2.1.4. Inferential Analysis

#### Confidence intervals:

When applicable, bilateral asymptotic or exact confidence intervals for binomial distributions will be calculated at the 95% level.

For categorical variables, if pertinent, the 95% asymptotic confidence interval will be calculated if theoretical assumptions are verified. If this is not the case, and the corresponding proportion is 0% or 100%, then the Agresti-Coull confidence interval will be calculated instead. In all other cases, the exact confidence interval will be calculated.

#### · Survival analysis:

Time-to-event variables will be described over time by survival curves as per the Kaplan-Meier method together with the associated estimators, considering the upper window of the corresponding visits. The survival rate will be presented at each time point (30 days, 90 days, 180 days, 365 days) and overall.

## 2.1.5. Data Listings

Patient data listings will be selected data supportive of summary statistical tables, including derived/calculated data from statistical process. These data listings are performed on selected analysis sets according to the focus of the analysis and are sorted by subject number and visit. Data entry into a free field in the CRF will be described in the listings.

### 2.2. Sample size calculation

Up to 60 subjects in total will be enrolled at up to four sites in this clinical safety and feasibility study. Approved sites will enroll at least 5 and not more than 30 subjects.

### 2.3. Analysis Sets

## 2.3.1. Definition of patient populations

3 populations will be defined:

- The enrolled population will include all subjects who provided their informed consent.
- Safety Subjects/Intent to Treat Subjects (ITT) population will include all enrolled subjects except those who terminate their participation prior to the beginning of the Index Procedure.
- The Per Protocol (PP) population will include Intent-to-treat subjects for whom the Index Procedure is finished without interfering investigational device deficiency or malfunction.

The primary feasibility endpoint will be analyzed on ITT and on PP population.



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


#### 2.3.2. Protocol Deviations

A description of the deviation from the protocol and justification must be recorded on the Protocol Deviation Form. The deviations are defined as follows:

- Consentement inappropriately obtained
- Procedure not performed according to protocol/IFU
- Inclusion/Exclusion Criteria deviation
- Protocol required test not completed
- Missed Follow-up visit
- Follow-up visit performed outside of window
- Other

#### 2.3.1. Databases

The Remapping at 60 Days, recurrence and Additional endpoints analysis will be based on the MDT Excel file sent by sponsor, which will contain:

- Received ablation at remap"
- Received RF/PFA ablation at remap
- Patient with Early recurrence of atrial fibrillation (AF)
- AF status at remapping procedure
- AF free survival days
- Atrial fibrillation/ Atrial flutter / Atrial tachycardia (AF/AFL/AT) status at remapping procedure
- AF/AFL/AT free survival days
- 6-month holter
- 12-month holter
- Transtelephonic monitor (TTM) weeks expected
- TTM weeks received
- Number TTM transmissions
- Radiofrequency (RF) touchup
- Ablation (ABL) >90 days Blanking period
- Class I/III antiarrhythmics drug (AAD) >90 days
- Amiodarone
- Direct current cardioversion (DCCV) >90 days
- Arrhythmia-related (AF, AFL, AT) hospitalization

The Excel file sent by the Sponsor will have the same structure (in terms of variables names, labels, formats) for each analysis to ensure the continuity of the programming.

Corelab data will be received, but no analysis will be done. All the data will be received in the MDT file from the sponsor

All other analysis will be done on the e-CRF clinical database.



FARAPULSE\_PersAFOne II SAP V1.0 PERSAFONE II V1.0


## 2.4. Statistical Analyses

## 2.4.1. Patient Disposition and Follow-up

## 2.4.1.1. Patient Populations Sample Size

The number and percentage of patients included in each population and the reasons of non-inclusion in each subsequent population will be presented on the enrolled population.

The number of patients included, as well as the distribution by center will be presented globally. The number and percentage of patients present at each visit will be presented with the study exit reasons.

A listing will be provided to present patient disposition. The following variables will be listed:

- Date of consent
- Procedure date
- Remap date
- Most recent follow-up
- Date of study exit
- Follow up time (days)

## 2.4.1.2. Protocol Deviations

Frequency of patients with at least one protocol deviation, as well as the total number of events, will be summarized on the ITT population, by Type of deviation.

The detail will be also presented in a listing.

#### 2.4.2. Baseline Patient Characteristics

Descriptive statistical data will be used to draw up a recapitulation of the characteristics of the patients at the time of enrolment. It will be summarized on the ITT population.

- Demographics at baseline: Age, Gender, height, weight, BMI
- Baseline Medical History: CHA2DS2-VASc Score, heart rate, blood pressure, Months between
  Date of first documented AF diagnosis and Enrollment date, number of AF episodes past year,
  Months between Date of most recent AF episode and Enrollment date, failed drug,
  Hypertension, Cardiac arrhythmias, CT/MRI results, Echocardiography, LVEF, Left Atrial AP
  Diameter, Hypertension

Previous parameters will also be presented in a listing.

#### 2.4.3. Index Procedure

Descriptive statistical data will be used to draw up a recapitulation of the intervention details at the time of the procedure.

The following data will be presented on the ITT population:

Procedure Data: Procedure time (hours), Farawave dwell total time (hours), PVI ablation time (hours), FARAPOINT CTI dwell TOTAL (hours), CTI Experimental ablation catheter time, Total fluoroscopy time (minutes), Total volume contrast (cc), Total Volume IV Fluids (cc); Total number of PVI ablations, Total number of ablations for each vein, Total number of PVI ablations by patient, PVI status at end of procedure by each attempted vein, Num PV treated, Num PV isolated, Proportion of veins isolated, CTI acute isolation, Total number of ablations of CTI applications, LA floor attempted and LA floor Isolated/Blocked, LA roof attempted and LA roof



FARAPULSE\_PersAFOne II SAP V1.0 PERSAFONE II V1.0


Isolated/Blocked, LA MI attempted and LA MI Isolated/Blocked, LAPW attempted and LAPW Isolated/Blocked, Total number of ablations for LAPW, Total number of ablations for LAPW with FARAWAVE, LAPW Experimental ablation catheter time,

A listing will be provided to present previous parameters.

## 2.4.4. Follow-up at remapping procedure

Descriptive statistical data will be used to draw up a recapitulation of the follow-up details at the remap procedure.

The following data will be presented on the ITT population:

Remapping details: Days follow up at remap, Durable PVI, LSPV chronic isolation, LIPV chronic isolation, LCPV chronic isolation, RSPV chronic isolation, RIPV chronic isolation, RMPV chronic isolation, CTI chronic isolation, LAPW chronic isolation, Number of veins durably isolated, Number of veins with gaps.

The details will also be presented in a listing.

## 2.4.5. 6 and 12 Months follow up

Descriptive statistical data will be used to draw up a recapitulation of the follow-up details at 6 and 12 Months follow up.

The following data will be presented on the ITT population:

TTM compliance and Holter compliance at 6 months and 12 months. Freedom from AF/AFL/AT (for patient On AADs and on patient Off AADs), Freedom from AF (for patient On AADs and on patient Off AADs), Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days (for patient On AADs and on patient Off AADs), Freedom from AF, no DCCV>90 days, no RF, no ablation >90 days (for patient On AADs and on patient Off AADs).

## 2.4.6. Feasibility Analysis

The feasibility analysis will be performed on the ITT population.

### 2.4.6.1. Primary Feasibility Analysis

The proportion of subjects that achieve Acute Procedural Success (APS) defined as the percutaneous endocardial creation of a complete, electrically isolating set of lesions around the ostia of the pulmonary veins (PVI) using the FARAPULSE Cardiac Ablation System Plus during the Index Procedure, as clinically assessed by entrance and/or exit block performed  $\geq$  20 minutes after the last PVI lesion is made.

#### 2.4.6.2. Secondary Feasibility Analysis

The secondary feasibility analyses are:

- The proportion of subjects who undergo the protocol-specified 60-Day Remapping Procedure and achieve Chronic Procedural Success (CPS) defined as persistent electrical isolation of all initially ablated pulmonary veins. Chronic Procedural Success will be subdivided by Index Procedure only CPS and Reablated CPS subjects.
- The proportion of attempted subjects that achieve Acute CTI Success, defined as the creation of bi-directional electrical block across the CTI using the investigational devices.
- Durability of the CTI and/or other extra-PV lesion set(s), when applicable. Durability is defined as unaltered integrity of each such lesion assessed at the Remapping Procedure.
- The proportion of subjects that achieve Therapeutic Success, defined as freedom from:
  - Post-Blanking Period through assessment: occurrence of AF, AFL or AT, or ablation for AF/AFL/AT using the study device
  - At any time: ablation for AF/AFL/AT with a non-study device



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


Therapeutic Success will be assessed from the end of the 90 Day Blanking Period through Months 6 and 12 and will be subdivided by on / off AFDs (Atrial Fibrillation Drugs) post-Blanking Period.

## 2.4.7. Additional endpoints

The additional observations will be performed on the ITT population and will include:

- Proportion of subjects with early recurrence of atrial fibrillation (ERAF) by 90 days after the initial study ablation.
- Time to Therapeutic Failure
- Proportion of all ablated pulmonary veins that are isolated at the Index Procedure using the study device.
- Proportion of all ablated pulmonary veins isolated using the study device during the Index Procedure that remain isolated at the 60-day Remapping Procedure.
- The proportion of attempted subjects that achieve Chronic CTI Success, defined as persistent bi-directional electrical block across the CTI as assessed at the 60-day remapping procedure.
- The proportion of attempted subjects that achieve Chronic Focal Success, defined as persistent electrical nonconductivity of extra-PV tissue targeted for ablation in the Index Procedure, excluding the CTI as assessed at the 60 day remapping procedure.

## 2.4.8. Safety Endpoint

Descriptive statistical data is used to analyze the Primary Safety Endpoint (PSE), the secondary safety endpoints and others analysis. The analysis is performed on the ITT populations.

The Safety endpoint will be performed on the ITT population and will include

### 2.4.8.1. Primary Safety Analysis

The primary safety endpoint for this study is the Composite Safety Endpoint (CSE) defined as the incidence of the following early-onset and late-onset serious adverse events (SAEs) which are device- or procedure-related, as adjudicated by the CEDMC.

Composite Safety Endpoint Definitions.

- Early onset (within 30 days of an Index or Remap Procedure)
  - Death
  - Myocardial infarction (MI)
  - Persistent diaphragmatic paralysis
  - Stroke or transient ischemic attack (TIA)
  - Peripheral or organ thromboembolism
  - Pericarditis
  - Cardiac tamponade / perforation
  - Vascular access complications requiring intervention
  - Heart block
- Late onset (any time during follow-up through 12 months)
  - Pulmonary vein (PV) stenosis (> 70% diameter reduction from baseline)
  - Atrio-esophageal fistula

#### 2.4.8.2. Secondary Safety Analysis

The Primary Safety Endpoint assessed at 7 rather than 30 days



FARAPULSE\_PersAFOne II SAP V1.0 PERSAFONE II

INOAI OINE II

V1.0


- The proportion of subjects with a device- or procedure-related SAE
- The proportion of subjects with stroke or TIA
- The proportion of subjects requiring cardioversion
- The proportion of subjects requiring an arrhythmia-related hospitalization

#### 2.4.9. Concomitant Medications

Concomitant medications will be listed on the ITT population.

#### 2.5. Derived Criteria Calculation

If at least one of the items needed to calculate a derived criteria is missing, then the corresponding derived criteria will be considered as missing.

#### Patient Disposition:

• Derived criteria "Enrolled population" will be derived as follows:

IF the date of patient consent is filled in **Patient eligibility form (IE) THEN** "Enrolled population" = 'Yes'

ELSE "Enrolled population" = 'No'.

• Derived criteria "ITT population" will be defined as follows:

**IF** "Enrolled population" = 'Yes' and the date of the Procedure is filled in **Procedural data form (PR) THEN** "ITT population" = 'Yes'

ELSE "ITT population" = 'No'.

• Derived criteria "Per Protocol population PP" will be defined as follows:

IF "ITT population" = 'Yes' AND Device Deficiency Number is not filled AND Serial # is not filled in **Device Deficiency DD Form THEN** Per Protocol population = 'Yes'

**ELSE** Per Protocol population = 'No'.

Derived criteria "Time of patient follow-up" will be calculated as:
 Date of study exit/withdrawal (\*) in Patient eligibility form (IE) – date of procedure in Procedural data form (PR)

\*if the patient is still in the study, the last visit date will be used instead of the exit/ withdrawal one.

- Derived criteria "Study exit by visit" will be calculated as:
  - IF STUDY EXIT DATE <PROCEDURE DATE THEN patient exited study Before Procedure.</p>
  - ELSE IF STUDY EXIT DATE≥PROCEDURE DATE AND (DISCHARGE DATE is missing AND 30 DAYS VISIT DATE is missing AND REMAP DATE is missing AND 6 MONTHS VISIT DATE is missing AND 12 MONTHS VISIT DATE is missing) THEN patient exited study after Procedure.
  - ELSE IF STUDY EXIT DATE > DISCHARGE DATE AND (30 DAYS VISIT DATE is missing AND REMAP DATE is missing AND 6 MONTHS VISIT DATE is missing AND 12 MONTHS VISIT DATE is missing) THEN patient exited study after Discharge.
  - ELSE IF STUDY EXIT DATE ≥ 30 DAYS VISIT DATE AND (REMAP DATE is missing AND 6 MONTHS VISIT DATE is missing AND 12 MONTHS VISIT DATE is missing) THEN patient exited study after 30 days visit.



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II


V1.0

- ELSE IF STUDY EXIT DATE≥ REMAP DATE AND (6 MONTHS VISIT DATE is missing AND 12 MONTHS VISIT DATE is missing) THEN patient exited study after Remap procedure.
- ELSE IF STUDY EXIT DATE ≥ 6 MONTHS VISIT DATE AND (12 MONTHS VISIT DATE is missing) THEN patient exited study after 6 months.
- ELSE ĬF STUDY EXIT DATE≥12 MONTHS VISIT DATE THEN patient exited study after 12 months.

#### **Baseline Patient Characteristics:**

- Derived criteria "Time between the first documented AF diagnosis and the enrollment (months)" will be defined as follows:
  - (Informed consent date date of first documented AF diagnosis) /30.4167 in **AF history form** (AH).
- Derived criteria "Time between the most recent AF episode and the enrollment (months)" will be defined as follows:
  - (Informed consent date date of most recent AF episode) /30.4167 in AF history form (AH).

#### Index Procedure:

- Derived criteria "Procedure time (hours)" will be defined as follows:
   Procedure end- Procedure start in Procedural data form (PR).
- Derived criteria "PVI ablation time (hours)" will be defined as follows:
   Last PVI ablation\* time First PVI ablation\* time in Procedural data form (AB)
- \*Where ablation location ablation location: ablation location = ("Left superior", "Left inferior", "Right superior", "Right inferior", "Left common ostium", "Right middle") and (Ablation location='Other" and Ablation location, Other specify='LCPV')).
- Derived criteria "FARAWAVE dwell time (hours)" will be defined as follows:
   SUM of [(FARAWAVE ablation catheter remove 1 FARAWAVE ablation catheter introduction 1), (FARAWAVE ablation catheter remove n FARAWAVE ablation catheter introduction n)] in Procedural data form (PR)
  - \* FARAWAVE ablation catheter remove/introduction = Ablation catheter remove/introduction WHERE FARAWAVE: Type of endocardial catheter used for ablation is Ticked OR Type of endocardial catheter used for ablation = 'FARAWAVE'
- Derived criteria "CTI (FARAPOINT) dwell time (hours)" will be defined as follows:
   SUM of [(FARAPOINT ablation catheter remove 1 FARAPOINT ablation catheter introduction 1),
  - (FARAPOINT ablation catheter remove n FARAPOINT ablation catheter introduction n)] in Procedural data form (PR)
  - \* FARAPOINT ablation catheter remove/introduction = Ablation catheter remove/introduction WHERE FARAPOINT: Type of endocardial catheter used for ablation is Ticked OR Type of endocardial catheter used for ablation = FARAPOINT
- Derived criteria "LAPW ablation time (hours)" will be defined as follows:
   Last LAPW ablation time First LAPW ablation time in Procedural data form (AB)



FARAPULSE\_PersAFOne II SAP V1.0 PERSAFONE II

V1.0


- Derived criteria "Total number of PVI applications" will be defined as follows:
   SUM of [(Count (Ablation location IN ("Left superior", "Left inferior", "Right superior", "Right inferior", "Right middle", "Left common ostium") OR (Ablation location='Other" AND Ablation location, Other specify='LCPV'))] in Procedural data form (AB)
- Derived criteria "Number of LAPW applications" will be defined as follows:
   SUM of [(Count (Ablation location='Other" AND Ablation location, Other specify IN ("LA PW", "LAPW", "LEFT ATRIAL POSTERIOR WALL")] in Procedural data form (AB)
- Derived criteria "Total number of CTI applications" will be defined as follows: SUM of [(Count (Ablation location=" CTI")] in **Procedural data form (AB)**
- Derived criteria "Total number of veins treated" will be defined as follows:
   COUNT of ["left superior", "left inferior", "left common ostium", "right middle", "right superior", "right inferior"] WHERE isolated/Blocked in ('Yes', 'No') in Procedural data form (PR)
- Derived criteria "Total number of veins isolated" will be defined as follows:
   SUM of [left superior, left inferior, left common ostium, right middle, right superior, right inferior]
   WHERE isolated/Blocked = 'Yes' in Procedural data form (PR)
- Derived criteria "Of the total number of veins treated, the number of veins isolated (Proportion of veins isolated)" will be defined as follows:
   Derived criteria "Total number of veins isolated"/ Derived criteria "Total number of veins treated"
- Derived criteria Proportion "CTI acute isolation" will be defined as follows:
   COUNT of [CTI isolated/Blocked='Yes' /CTI Attempted='Yes'] in Procedural data form (PR)

#### Remapping at 60 Days

- Derived criteria "Days of follow-up at remapping procedure" will be defined as follows:
   Assessment date (WHERE Visit='60-Day Follow-up')' in Follow-up form (FU) Procedure date in Procedural data form (AB)
- Derived criteria "Durable PVI" will be defined as follows:

IF Any PV reconnection noted? = 'No' in Follow-up 3D electroanatomical mapping form (RM)
THEN PVI durable = 'Yes'

**ELSE IF** Any PV reconnection noted? = 'Yes' in **Follow-up 3D electroanatomical mapping form (RM) THEN** PVI Durable=No

- Derived criteria "LAPW chronic isolation" will be defined as follows:
  IF Anatomical Structure/Area other specification 1 IN ("POSTERIOR WALL" "LA POSTERIOR WALL" "LAPW" "PA WALL" "BOX POSTERIOR WALL") AND Other 1 Lesion durable = 'yes' OR Anatomical Structure/Area other specification 2 IN ("POSTERIOR WALL" "LA POSTERIOR WALL" "LAPW" "PA WALL" "BOX POSTERIOR WALL") AND Other 2 Lesion durable = ='Yes' in Follow-up 3D electroanatomical mapping form (RM) THEN LAPW chronic isolation= 'Yes' ELSE LAPW chronic isolation = 'No'
- Derived criteria "Num veins with isolation" will be defined as follows:



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


SUM OF [ (Anatomical structure/Area Isolated = ('Left superior, left inferior, Left common ostium, right superior, right inferior, right middle) AND Isolated (Yes/No/'N/A') ='Yes'] in Follow-up 3D electro anatomical mapping form (RM)

- Derived criteria "Num veins with gaps" will be defined as follows:
   SUM OF [ (Anatomical structure/Area Isolated = ('Left superior, left inferior, Left common ostium, right superior, right inferior) AND Isolated (Yes/No/'N/A') ='No'] in Follow-up 3D electro anatomical mapping form (RM)
- Derived criteria "Percentage of PVs Isolated per-vein at remap" will be defined as follows: (Num veins with isolation /(Num veins with isolation + Num veins with gaps))\*100
- Derived criteria "Num veins remain isolated" will be defined as follows:
   Derived criteria "Num PV isolated" Derived criteria "Num veins with gaps"
- Derived criteria "Proportion PVs Remaining isolated" will be defined as follows:
   Derived criteria "Num veins remain isolated" /Derived criteria "Num PV isolated"

#### 6 and 12 Months follow up

- Derived criteria "TTM compliance (%) (calculated)" will be defined as follows:
   (TTM weeks received /TTM weeks expected) \*100 in MDT excel file
- Derived criteria "Holter compliance (%) at 6 months" will be defined as follows:
   IF 6mo Holter in ('AF', 'none', 'SVT') in MDT excel file THEN Holter compliance (%) at 6 months = 'Yes'
  - ELSE IF 6mo Holter in ('MISSING') in **MDT excel file THEN** Holter compliance (%) at 6 months='No'
- Derived criteria "Holter compliance (%) at 12 months" will be defined as follows:
   IF 12mo Holter in ('AF', 'none', 'SVT') in MDT excel file THEN Holter compliance (%) at 12 months = 'Yes'
  - **ELSE IF** 12mo Holter in ('MISSING') in **MDT excel file THEN** Holter compliance (%) at 12 months='No'
- Derived criteria "Freedom from AF/AFL/AT" will be defined as follows:
   IF AF/AFL/AT status =0 in MDT excel file THEN Freedom from AF/AFL/AT ='Yes'
   ELSE Freedom from AF/AFL/AT ='No'
- Derived criteria "Freedom from AF/AFL/AT with Class I/III AAD >90 days" will be defined as follows:
  - IF AF/AFL/AT status =0 AND Class I/III AAD >90 days =1 in MDT excel file THEN Freedom from AF/AFL/AT with Class I/III AAD >90 days ='Yes'
  - ELSE Freedom from AF/AFL/AT with Class I/III AAD >90 days ='No'
- Derived criteria "Freedom from AF/AFL/AT without Class I/III AAD >90 days" will be defined as follows:



FARAPULSE\_PersAFOne II SAP

PERSAFONE II

V1.0


IF AF/AFL/AT status =0 AND Class I/III AAD >90 days =0 in MDT excel file THEN Freedom from AF/AFL/AT without Class I/III AAD >90 days = 'Yes'

ELSE Freedom from AF/AFL/AT without Class I/III AAD >90 days ='No'

- Derived criteria "Freedom from AF" will be defined as follows:
   IF AF status =0 in MDT excel file THEN Freedom from AF ='Yes'
   ELSE Freedom from AF ='No'
- Derived criteria "Freedom from AF with Class I/III AAD >90 days" will be defined as follows:
   IF AF status =0 AND Class I/III AAD >90 days =1 in MDT excel file THEN Freedom from AF with Class I/III AAD >90 days ='Yes'
  - ELSE Freedom from AF with Class I/III AAD >90 days ='No'
- Derived criteria "Freedom from AF without Class I/III AAD >90 days" will be defined as follows:
   IF AF status =0 AND Class I/III AAD >90 days =0 in MDT excel file THEN Freedom from AF without Class I/III AAD >90 days ='Yes'
  - ELSE Freedom from AF without Class I/III AAD >90 days ='No'
- Derived criteria "Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days" will be defined as follows:
  - **IF** AF/AFL/AT status =0 **AND** DCCV90D=0 **AND** RF touch up=0 **AND** ABL>90 day=0 in **MDT excel file THEN** Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days ='Yes'
  - ELSE Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days ='No'
- Derived criteria "Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days with Class I/III AAD >90 days" will be defined as follows:
  - IF AF/AFL/AT status =0 AND DCCV90D=0 AND RF touch up=0 AND ABL>90 day=0 AND Class I/III AAD >90 days =1 in MDT excel file THEN Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days with Class I/III AAD >90 days='Yes'
  - ELSE Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days with Class I/III AAD >90 days='No'
- Derived criteria "Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days without Class I/III AAD >90 days" will be defined as follows:
  - IF AF/AFL/AT status =0 AND DCCV90D=0 AND RF touch up=0 AND ABL>90 day=0 AND Class I/III AAD >90 days =0 in MDT excel file THEN Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days without Class I/III AAD >90 days= 'Yes'
  - ELSE Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days without Class I/III AAD >90 days='No'
- Derived criteria "Freedom from AF, no DCCV>90 days, no RF, no ablation >90 days" will be defined as follows:
  - IF AF status =0 AND DCCV90D=0 AND RF touch up=0 AND ABL>90 day=0 in MDT excel file THEN Freedom from AF, no DCCV>90 days, no RF, no ablation >90 days ='Yes' ELSE Freedom from AF, no DCCV>90 days, no RF, no ablation >90 days ='No'



FARAPULSE\_PersAFOne II SAP

PERSAFONE II


V1.0

 Derived criteria "Freedom from AF, no DCCV>90 days, no RF, no ablation >90 days with Class I/III AAD >90 days" will be defined as follows:

IF AF status =0 AND DCCV90D=0 AND RF touch up=0 AND ABL>90 day=0 AND Class I/III AAD >90 days =1 in MDT excel file THEN Freedom from AF, no DCCV>90 days, no RF, no ablation >90 days with Class I/III AAD >90 days ='Yes'

ELSE Freedom from AF, no DCCV>90 days, no RF, no ablation >90 days with Class I/III AAD >90 days ='No'

• Derived criteria "Freedom from AF, no DCCV>90 days, no RF, no ablation >90 days without Class I/III AAD >90 days" will be defined as follows:

IF AF status =0 AND DCCV90D=0 AND RF touch up=0 AND ABL>90 day=0 AND Class I/III AAD >90 days =0 in MDT excel file THEN Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days without Class I/III AAD >90 days='Yes'

ELSE Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days without Class I/III AAD >90 days= 'No'

#### Primary Feasibility endpoint

Derived criteria "Acute Procedural Success (APS)" will be defined as follows
 IF Ablation with study device was successful = 'Yes' in procedural form (PR) THEN APS='Yes'
 ELSE IF Ablation with study device was successful = 'No' in procedural form (PR) THEN APS='No'

#### Secondary Feasibility endpoint

• Derived criteria "Chronic Procedural Success (CPS)" will be defined as follows:

IF Has all ablation with the study device(s) been successful? ='Yes' in **Procedural data form** (**PR)** AND Has all ablation with the study device remain successful? ='Yes' AND Additional ablation(s) performed? ='No' in **FOLLOW UP 3D ELECTRO ANATOMICAL MAPPING form** (**RM)** THEN Chronic Procedural Success (CPS) ='Yes, index procedure only'

**ELSE IF** Has all ablation with the study device(s) been successful? ='Yes' in **Procedural data form (PR) AND** Has all ablation with the study device remain successful? ='No' **AND** Any PV reconnections noted? in **= 'Yes' AND** Additional ablation(s) performed? ='Yes' in **FOLLOW UP 3D ELECTRO ANATOMICAL MAPPING form (RM) THEN** Chronic Procedural Success (CPS) ='Yes, reblated'

**ELSE IF** Has all ablation with the study device(s) been successful? ='No' in **Procedural data** form (PR) THEN Chronic Procedural Success (CPS) ='No'

- Derived criteria "Acute CTI Success" will be defined as follows:
   COUNT of [CTI isolated/Blocked='Yes'/ CTI Attempted='Yes'] in Procedural data form (PR)
- Derived criteria "Durability of CTI at remap," will be defined as follows:
  - IF CTI lesion durable ='Yes' in Follow-up 3D electroanatomical mapping form (RM) THEN Durability of CTI at remap = 'Yes'
  - ELSE IF CTI lesion durable ='No' in Follow-up 3D electroanatomical mapping form (RM) THEN Durability of CTI at remap = 'No'
- Derived criteria "Durability of Mitral isthmus at remap" will be defined as follows:
  - IF Mitral isthmus lesion durable ='Yes' in Follow-up 3D electroanatomical mapping form (RM) THEN Durability of Mitral isthmus at remap = 'Yes'

**ELSE IF** Mitral isthmus lesion durable ='No' in **Follow-up 3D electroanatomical mapping form (RM) THEN** Durability of Mitral isthmus at remap = 'No'



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II


V1.0

Derived criteria "Durability of Left atrial roof line at remap" will be defined as follows:
 IF Left atrial roof line lesion durable ='Yes' in Follow-up 3D electroanatomical mapping form (RM) THEN Durability of Left atrial roof line at remap = 'Yes'
 ELSE IF Left atrial roof line lesion durable ='No' in Follow-up 3D electroanatomical mapping form (RM) THEN Durability of Left atrial roof line at remap = 'No'

- Derived criteria "Durability of Left atrial Posterior line" will be defined as follows:
   IF Left atrial Posterior line lesion durable ='Yes' in Follow-up 3D electroanatomical mapping form (RM) THEN Durability of Left atrial Posterior line at remap = 'Yes'
   ELSE IF Left atrial Posterior line lesion durable ='No' in Follow-up 3D electroanatomical mapping form (RM) THEN Durability of Left atrial Posterior line at remap = 'No'
  - Derived criteria "Durability of Left atrial Posterior wall" will be defined as follows:
- IF Anatomical Structure/Area other specification 1 IN ("POSTERIOR WALL" "LA POSTERIOR WALL" "LAPW" "PA WALL" "BOX POSTERIOR WALL") AND Other 1 Lesion durable = 'yes' OR Anatomical Structure/Area other specification 2 IN ("POSTERIOR WALL" "LA POSTERIOR WALL" "LAPW" "PA WALL" "BOX POSTERIOR WALL") AND Other 2 Lesion durable = 'Yes' in Follow-up 3D electroanatomical mapping form (RM) THEN LAPW chronic isolation= 'Yes'
- ELSE LAPW chronic isolation = 'No'
- Derived criteria "Therapeutic Success ON/OFF AAD" will be defined as follows:
   IF "AF/AFL/AT status"= 0 AND "RF touchup"= 0 AND "ABL >90 days" = 0 in MDT excel file THEN therapeutic success='Yes'
   ELSE therapeutic success='No'
- Derived criteria "Therapeutic Success Off ADD" will be defined as follows:
   IF Therapeutic success =Yes' AND Class I/III AAD>90days=0 in MDT excel file THEN therapeutic success Off ADD ='YES'
   ELSE IF Therapeutic success ='No' AND Class I/III AAD>90days=0 in MDT excel file THEN THEN therapeutic success Off ADD ='NO'
- Derived criteria "Therapeutic Success On ADD" will be defined as follows:
   IF Therapeutic success = 'Yes' AND Class I/III AAD>90days=1 in MDT excel file THEN therapeutic success On ADD = 'No'
   Else IF Therapeutic success = 'No' AND Class I/III AAD>90days=1 in MDT excel file THEN THEN therapeutic success On ADD = 'No'

#### Additional endpoints

 Derived criteria "Proportion of all ablated pulmonary veins that are isolated at the Index Procedure using the study device" will be defined as follows:

COUNT of [(Left Superior Isolated/Blocked ='Yes', Left Inferior Isolated/Blocked='Yes', Left Common Ostium Isolated/Blocked='Yes', Right Middle Isolated/Blocked='Yes', Right Superior Isolated/Blocked='Yes', Right Inferior Isolated/Blocked='Yes')] / COUNT of [(Left Superior Isolated/Blocked in (Yes, No), Left Common Ostium Isolated/Blocked in (Yes, No), Right Middle Isolated/Blocked in (Yes, No), Right Superior



form (PR)

# STATISTICAL ANALYSIS PLAN

FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0

Isolated/Blocked in (Yes, No), Right Inferior Isolated/Blocked in (Yes, No))] in **Procedural data** 

 Derived criteria "Proportion of all ablated pulmonary veins isolated using the study device during the Index Procedure that remain isolated at the 60-day remapping procedure" will be defined as follows:

(Derived criteria "Total number of veins isolated" - Derived criteria "Number of veins with gaps")/ Derived criteria "Total number of veins isolated"

• Derived criteria Proportion "Chronic CTI at 60d remap" will be defined as follows:

IF CTI lesion durable ='Yes' in Follow-up 3D electroanatomical mapping form (RM) THEN Chronic CTI at 60d remap ='Yes'

ELSE IF CTI lesion durable ='No' in Follow-up 3D electroanatomical mapping form (RM) THEN Chronic CTI at 60d remap ='No'

Derived criteria "Chronic Focal Success" will be defined as follows:
 IF Anatomical Structure/Area other specification 1 IN ("POSTERIOR WALL" "LA POSTERIOR WALL" "POSTERIOR WALL" "POSTERIOR WALL" "POSTERIOR WALL" "POSTERIOR WALL" "LA POSTERIOR WALL" "LA POSTERIOR WALL" "LA POSTERIOR WALL" "LAPW" "PA WALL" "BOX POSTERIOR WALL") AND Other 2 Lesion durable = "Yes' in Follow-up 3D electroanatomical mapping form (RM) THEN Chronic focal success "Yes'

#### Primary Safety endpoint

ELSE Chronic focal succes = 'No'

Unless otherwise indicated, all the following variables will be derived from the Adverse event adjudication form (CE)

Derived criteria "Death" will be defined as follows:

IF (30≤ (EVENT DATE-PROCEDURE DATE IN PROCEDURAL DATA FORM (PR)) OR (30≤ (EVENT DATE-≤REMAPPING DATE IN FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' Death' THEN DEATH='Yes'

**ELSE DEATH='No'** 

Derived criteria "Myocardial infarction" will be defined as follows:

IF (30≤ (EVENT DATE-PROCEDURE DATE IN PROCEDURAL DATA FORM (PR)) OR (30≤ (EVENT DATE-REMAPPING DATE IN FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' Myocardial infarction' THEN Myocardial infarction='Yes'.

**ELSE** Myocardial infarction ='No'.

Derived criteria "PV Stenosis" will be defined as follows:

IF (0≤ (EVENT DATE-PROCEDURE DATE IN **PROCEDURAL DATA FORM (PR)**) ≤360 **AND** PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' PV Stenosis' **THEN** PV Stenosis ='Yes'. **ELSE** PV Stenosis ='No'.



FARAPULSE\_PersAFOne II SAP

PERSAFONE II

V1.0


• Derived criteria "Diaphragmatic Paralysis" will be defined as follows:

IF (30≤ (EVENT DATE-PROCEDURE DATE IN PROCEDURAL DATA FORM (PR)) OR (30≤ (EVENT DATE-REMAPPING DATE IN FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' Diaphragmatic Paralysis' THEN Diaphragmatic Paralysis ='Yes'.

**ELSE** Diaphragmatic Paralysis ='No'.

Derived criteria "AE fistula" will be defined as follows:

IF (0≤ (EVENT DATE-PROCEDURE DATE IN **PROCEDURAL DATA FORM (PR)**) ≤360 **AND** PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' AE fistula' **THEN** AE fistula ='Yes'. **ELSE** AE fistula ='No'.

• Derived criteria "TIA" will be defined as follows:

IF (30≤ (EVENT DATE-PROCEDURE DATE IN PROCEDURAL DATA FORM (PR)) OR (30≤ (EVENT DATE-REMAPPING DATE IN FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' TIA' THEN TIA=Yes. ELSE TIA='No'.

Derived criteria "CVA" will be defined as follows:

IF (30≤ (EVENT DATE-PROCEDURE DATE IN **PROCEDURAL DATA FORM (PR)) OR** (30≤ (EVENT DATE-REMAPPING DATE IN **FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)**) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' CVA' THEN CVA='Yes'. ELSE CVA='No'.

• Derived criteria "Major pericarditis" will be defined as follows:

IF (30≤ (EVENT DATE-PROCEDURE DATE IN PROCEDURAL DATA FORM (PR)) OR (30≤ (EVENT DATE-REMAPPING DATE IN FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' Major pericarditis' THEN Major pericarditis = 'Yes'.

ELSE Major pericarditis ='No'.

Derived criteria "Tamponade/Perforation" will be defined as follows:

IF (30≤ (EVENT DATE-PROCEDURE DATE IN PROCEDURAL DATA FORM (PR)) OR (30≤ (EVENT DATE-REMAPPING DATE IN FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' Tamponade/Perforation' THEN Tamponade/Perforation ='Yes'

ELSE Tamponade/Perforation ='No'.

Derived criteria "Heart Block" will be defined as follows:

IF (30≤ (EVENT DATE-PROCEDURE DATE IN PROCEDURAL DATA FORM (PR)) OR (30≤ (EVENT DATE-REMAPPING DATE IN FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' Heart Block' THEN Heart Block ='Yes'

ELSE Heart Block ='No'



FARAPULSE\_PersAFOne II SAP

PERSAFONE II

V1.0


Derived criteria "Vascular Access Complication" will be defined as follows:
 IF (30≤ (EVENT DATE-PROCEDURE DATE IN PROCEDURAL DATA FORM (PR)) OR (30≤ (EVENT DATE-REMAPPING DATE IN FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' Vascular Access Complication' THEN Vascular Access Complication ='Yes'

**ELSE** Vascular Access Complication ='No'

 Derived criteria "Total Early and Late Onset Composite Safety Endpoint" will be defined as follows:

IF Death=Yes OR Myocardial infarction =Yes OR PV Stenosis =Yes OR Diaphragmatic Paralysis =Yes OR AE fistula =Yes OR TIA =Yes OR CVA=Yes OR Major pericarditis =Yes OR Tamponade/Perforation =Yes OR Heart Block =Yes OR Vascular Access Complication =Yes THEN Total Early and Late Onset Composite Safety Endpoint ='Yes'

ELSE Total Early and Late Onset Composite Safety Endpoint ='No'

Derived criteria "Total Early Onset Composite Safety Endpoint" will be defined as follows:
 IF Death=Yes OR Myocardial infarction =Yes OR Diaphragmatic Paralysis =Yes OR TIA =Yes
 OR CVA=Yes OR Major pericarditis =Yes OR Tamponade/Perforation =Yes OR Heart Block
 =Yes OR Vascular Access Complication =Yes THEN Total Early Onset Composite Safety Endpoint='Yes'

ELSE Total Early Onset Composite Safety Endpoint='No'

 Derived criteria "Total Late (any time during follow-up through 12 months)" will be defined as follows:

IF PV Stenosis =Yes OR AE fistula =Yes THEN Total Late (any time during follow-up through 12 months) ='Yes'

ELSE Total Late (any time during follow-up through 12 months) ='No.

#### Secondary Safety endpoint

Unless otherwise indicated, all the following variables will be derived from the Adverse event adjudication form (CE)

• Derived criteria "Death 7 days" will be defined as follows:

IF (7≤ (EVENT DATE-PROCEDURE DATE IN PROCEDURAL DATA FORM (PR)) OR (7≤ (EVENT DATE-REMAPPING DATE IN FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' Death' THEN DEATH='Yes'

**ELSE DEATH='No'** 

Derived criteria "Myocardial infarction 7 days" will be defined as follows:

IF (7≤ (EVENT DATE-PROCEDURE DATE IN **PROCEDURAL DATA FORM (PR)) OR** (7≤ (EVENT DATE-REMAPPING DATE IN **FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)**) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' Myocardial infarction' THEN Myocardial infarction='Yes'.

**ELSE** Myocardial infarction = 'No'.

Derived criteria "Diaphragmatic Paralysis 7 days" will be defined as follows:

IF ( $7 \le$  (EVENT DATE-PROCEDURE DATE IN **PROCEDURAL DATA FORM (PR)**) OR ( $7 \le$  (EVENT DATE-REMAPPING DATE IN **FOLLOW-UP 3D ELECTROANATOMICAL MAPPING** 



FARAPULSE\_PersAFOne II SAP

PERSAFONE II

V1.0


**FORM (RM)** ) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' Diaphragmatic Paralysis' THEN Diaphragmatic Paralysis ='Yes'.

**ELSE** Diaphragmatic Paralysis = 'No'.

Derived criteria "TIA 7 days" will be defined as follows:
 IF (7≤ (EVENT DATE-PROCEDURE DATE IN PROCEDURAL DATA FORM (PR)) OR (7≤ (EVENT DATE-REMAPPING DATE IN FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' TIA' THEN TIA='Yes'.
 ELSE TIA='No'.

Derived criteria "CVA 7 days" will be defined as follows:
 IF (7≤ (EVENT DATE-PROCEDURE DATE IN PROCEDURAL DATA FORM (PR)) OR (7≤ (EVENT DATE-REMAPPING DATE IN FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' CVA' THEN CVA='Yes'. ELSE CVA='No'.

Derived criteria "Major pericarditis 7 days" will be defined as follows:

IF (7≤ (EVENT DATE-PROCEDURE DATE IN **PROCEDURAL DATA FORM (PR)) OR** (7≤ (EVENT DATE- REMAPPING DATE IN **FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)**) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' Major pericarditis' THEN Major pericarditis = 'Yes'.

**ELSE** Major pericarditis = 'No'.

• Derived criteria "Tamponade/Perforation 7 days" will be defined as follows:

IF (7≤ (EVENT DATE-PROCEDURE DATE IN PROCEDURAL DATA FORM (PR)) OR (7≤ (EVENT DATE-REMAPPING DATE IN FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' Tamponade/Perforation' THEN Tamponade/Perforation = 'Yes'.

**ELSE** Tamponade/Perforation = 'No'.

Derived criteria "Heart Block 7 days" will be defined as follows:

IF (7≤ (EVENT DATE-PROCEDURE DATE IN PROCEDURAL DATA FORM (PR)) OR (7≤ (EVENT DATE-REMAPPING DATE IN FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' Heart Block' THEN Heart Block = 'Yes'.

**ELSE** Heart Block = 'No'.

Derived criteria "Vascular Access Complication 7 days" will be defined as follows:
 IF (7≤ (EVENT DATE-PROCEDURE DATE IN PROCEDURAL DATA FORM (PR)) OR (7≤ (EVENT DATE-REMAPPING DATE IN FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM)) AND PRIMARY SAFETY ENDPOINT EVENT CRITERIA=' Vascular Access Complication' THEN Vascular Access Complication = 'Yes'.

ELSE Vascular Access Complication = 'No'.

 Derived criteria "Total Early Onset Composite Safety Endpoint assessed at 7 days" will be defined as follows:

IF Death 7 days='Yes' OR Myocardial infarction 7 days='Yes' OR Diaphragmatic Paralysis 7 days='Yes' OR TIA 7 days='Yes' OR CVA 7 days='Yes' OR Major pericarditis 7 days='Yes' OR



FARAPULSE\_PersAFOne II SAP

PERSAFONE II

V1.0


Tamponade/Perforation 7 days='Yes' OR Heart Block 7 days='Yes' OR Vascular Access Complication 7 days='Yes' THEN Total Early Onset Composite Safety Endpoint assessed at 7 days = 'Yes'.

ELSE Total Early Onset Composite Safety Endpoint assessed at 7 days = 'No'.

- Derived criteria "Device-Related Serious Adverse Events (SAEs)" will be defined as follows:
   IF CEC seriousness = "Serious" AND CEC relationship to study Device in (Causal relationship, Probably related, Possibly related, Unlikely to be related) in adverse event adjudication form THEN Device-Related Serious Adverse Events (SAEs)='Yes'; ELSE Device-Related Serious Adverse Events (SAEs)='No'
- Derived criteria "Procedure-Related Serious Adverse Events (SAEs)" will be defined as follows:
   IF CEC relationship to study procedure in (Causal relationship, Probably related, Possibly related, Unlikely to be related) AND CEC seriousness = "Serious" THEN Procedure-Related Serious Adverse Events (SAEs)="Yes"
  - **ELSE IF** CEC relationship to study procedure ='Not related' **AND** CEC seriousness =" Serious" **THEN** Procedure-Related Serious Adverse Events (SAEs)='No'
- Derived criteria "Cardioversion" will be defined as follows:
  - IF Arrythmia-Treatment DC Cardioversion is ticked in **Arrythmia episodes form THEN** Cardioversion ='Yes';
  - **ELSE** Cardioversion ='No'
- Derived criteria "Stroke after index procedure" will be defined as follows:

   The state of the state
  - IF Event name='STROKE' in Adverse event form AND Event start date ≥ Procedure date in Procedural data Form (PR) THEN STROKE='Yes'
  - ELSE STROKE='No'
- Derived criteria "Transient Ischemic Attack (TIA) after index procedure" will be defined as follows:
   IF Event name=' Transient Ischemic Attack' in Adverse event form AND Event start date ≥
   Procedure date in Procedural data Form (PR) THEN TIA='Yes'
   ELSE TIA='No'
- Derived criteria "Stroke after Remap procedure" will be defined as follows:
   IF Event name='STROKE' in Adverse event form AND Event start date ≥ Remap date IN FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM) THEN STROKE='Yes' ELSE STROKE='No'
- Derived criteria "Transient Ischemic Attack (TIA) after Remap procedure" will be defined as follows:
  - IF Event name=' Transient Ischemic Attack' in Adverse event form AND Event start date ≥ Remap date in FOLLOW-UP 3D ELECTROANATOMICAL MAPPING FORM (RM) THEN TIA='Yes'
  - ELSE TIA='No'
- Derived criteria "Arrhythmia-related (AF, AFL, AT) hospitalization" will be defined as follows:
   IF Arrhythmia-related (AF, AFL, AT) hospitalization ='Yes' in MDT excel file THEN Arrhythmia-related (AF, AFL, AT) hospitalization ='Yes'
  - **ELSE IF** Arrhythmia-related (AF, AFL, AT) hospitalization ='No' in **MDT excel file THEN** Arrhythmia-related (AF, AFL, AT) hospitalization ='No'



FARAPULSE\_PersAFOne II SAP V1.0 PERSAFONE II V1.0 Page 26 /42

• Derived criteria "Death" will be defined as follows:

IF SAE: Death='Yes' in **Adverse event form OR** Reason ='Patient death' in **study exit form** THEN Death='Yes'

**ELSE** Death='No'

## 3. STATISTICAL SOFTWARE

All statistical outputs (summary tables and data listings) will be generated using SAS® version 9.4 or further.

# 4. STATISTICAL TABLES, LISTINGS AND GRAPHS (TABLE OF CONTENTS)

### 4.1. Statistical Tables

## 4.1.1. Table 1. Subject enrollment per Site

| | | Enrolled patients | ITT patients | PP patients |
|--------|-----------|-------------------|--------------|-------------|
| | | (N=XX) | (N=XX) | (N=XX) |
| Site # | Site Name | | | |
| XX | | XX (XX%) | XX (XX%) | XX (XX%) |
| XX | | XX (XX%) | XX (XX%) | XX (XX%) |

# 4.1.2. Table 2. Demographics

| | ITT Population | |
|---------|------------------------|-----------|
| | N = | XX |
| | Mean±S.D. | |
| | Median | [95% CI] |
| | (min, max)<br>(Q1, Q3) | [5570 C1] |
| | XX±X | |
| Age | XX | [XX - XX] |
| rige | (XX, XX) | |
| | (XX, XX) | |
| | $XX\pm X$ | |
| Height | XX | [XX - XX] |
| Tio giv | (XX, XX) | [121 121] |
| | (XX, XX) | |
| | XX±X | |
| Weight | XX | [XX - XX] |
| | (XX, XX) | [121 121] |
| | (XX, XX) | |
| BMI | XX±X | [XX - XX] |



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


| | (XX, XX)<br>(XX, XX) | |
|---------------|----------------------|-------------|
| | n/N (%) | [95% CI] |
| Male Gender | XX/XX (XX.X%) | [XX% - XX%] |
| Female Gender | XX/XX (XX.X%) | [XX - XX%] |

# 4.1.3. Table 3. Baseline Medical History

| | ITT Population<br>N = XX | |
|---|---|---|
| | Mean±S.D. Median (min, max) (Q1, Q3) | [95% CI] |
| Left atrial diameter (cm) | XX±X<br>XX<br>(XX, XX)<br>(XX, XX) | [XX - XX] |
| AF history (number of months between Date of first documented AF diagnosis and Enrollment date) | XX±X<br>XX<br>(XX, XX)<br>(XX, XX) | [XX - XX] |
| Number of AF episodes past year | XX±X<br>XX<br>(XX, XX)<br>(XX, XX) | [XX - XX] |
| AF history (number of between date of most recent AF episode and Enrollment dat) | XX±X<br>XX<br>(XX, XX)<br>(XX, XX) | [XX - XX] |
| Heart rate | XX±X<br>XX<br>(XX, XX)<br>(XX, XX) | [XX - XX] |
| Blood pressure | XX±X<br>XX<br>(XX, XX)<br>(XX, XX) | [XX - XX] |
| LVEF (%) | XX±X<br>XX<br>(XX, XX)<br>(XX, XX) | [XX - XX] |
| CHA2DS2VASC | XX±X<br>XX<br>(XX, XX) | [XX - XX] |



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


| | (XX, XX) | |
|------------------------------------------|------------------|-------------|
| | n/N (%) | [95% CI] |
| Patient that failed any AAD | XX/XX<br>(XX.X%) | [XX% - XX%] |
| If Yes: Class I | XX/XX<br>(XX.X%) | [XX% - XX%] |
| If Yes: Beta Blocker/Class II | XX/XX<br>(XX.X%) | [XX% - XX%] |
| If Yes: Class III | XX/XX<br>(XX.X%) | [XX% - XX%] |
| If Yes: Calcium Channel Blocker/Class IV | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Hypertension | XX/XX<br>(XX.X%) | [XX% - XX%] |
| CT/MRI results | , | |
| Left Superior Pulmonary Vein: Result | | |
| Normal | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Not Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Left Inferior Pulmonary Vein: Result | | |
| Normal | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Not Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Right Superior Pulmonary Vein: Result | | |
| Normal | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Not Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Right Inferior Pulmonary Vein: Result | | |
| Normal | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Not Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Mitral Valve: Result | | |



FARAPULSE\_PersAFOne II SAP PERSAFONE II V1.0 Page 29 /42

| Normal | XX/XX<br>(XX.X%) | [XX% - XX%] |
|---|---|---|
| Abnormal Not Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Left Ventricule: Result | | |
| Normal | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Not Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Right Atrium: Result | | |
| Normal | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Not Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Other finding 1: Result | | |
| Normal | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Not Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Other finding 2: Result | | |
| Normal | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Not Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Abnormal Clinically Significant | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Echocardiography | | |
| Protocol-required imaging for exclusion of LA thrombus performed | | |
| Yes | XX/XX<br>(XX.X%) | [XX% - XX%] |
| No | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Thrombus present | | |
| Yes | XX/XX<br>(XX.X%) | [XX% - XX%] |
| No | XX/XX | [XX% - XX%] |



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


| Ī | (XX.X%) |
|---|---------|
| | \ |

## 4.1.4. Table 4. Procedure

| | ITT Population | |
|----------------------------------|----------------------|-------------|
| | N = XX | |
| | Mean±S.D. | |
| | Median | [95% CI] |
| | $(\min, \max)$ | [, , , , ,] |
| | (Q1, Q3) | |
| | XX±X | |
| | XX | [XX - XX] |
| Procedure time (hours) | (XX, XX)<br>(XX, XX) | |
| Frocedure time (nours) | XX±X | |
| | XX | |
| | (XX, XX) | [XX - XX] |
| FARAWAVE dwell time (hours) | (XX, XX) | |
| Thu thit E are time (notice) | XX±X | |
| | XX | |
| | (XX, XX) | [XX - XX] |
| PVI ablation time (hours) | (XX, XX) | |
| , , | XX±X | |
| | XX | FX7X7 X7X7 |
| | (XX, XX) | [XX - XX] |
| FARAPOINT CTI dwell time (hours) | (XX, XX) | |
| | XX±X | |
| | XX | [XX - XX] |
| | (XX, XX) | |
| LAPW ablation time (hours) | (XX, XX) | |
| | XX±X | |
| | XX | [XX - XX] |
| | (XX, XX) | |
| Fluoroscopy time (min) | (XX, XX) | |
| | XX±X | |
| | XX | [XX - XX] |
| Contract values (co) | (XX, XX) | |
| Contrast volume (cc) | (XX, XX) | |
| | XX±X | |
| | XX | [XX - XX] |
| IV fluid volume (cc) | (XX, XX)<br>(XX, XX) | |
| · | ` ´ | NT A |
| Total number of PVI applications | XX | NA |
| Number of amlianticas/actions | XX±X | [XX - XX] |
| Number of applications/patient | XX | |



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


| | (XX, XX)<br>(XX, XX) | |
|---|---|---|
| Number of applications/vein | XX | NA |
| Number of LAPW applications | XX | NA |
| | N, n, n/N (%) | 95% CI |
| Total number of veins treated | XX | NA |
| Total number of veins isolated | XX | NA |
| Of the total number of veins treated, the number of veins isolated | XX/XX<br>(XX.X%) | [XX% - XX%] |
| CTI acute isolation | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Total number of CTI applications | XX | NA |

# 4.1.5. Table 5. Remap at 60 Days

| | | ITT Population $N = 25$ |
|---|---|---|
| | Mean±S.D. | |
| | Median | [95% CI] |
| | (min, max) | [9370 CI] |
| | (Q1, Q3) | |
| | $XX\pm X$ | |
| Days follow up at remap | XX | [XX - XX] |
| Buys follow up at follow | (XX, XX) | |
| | (XX, XX) | |
| | n/N (%) | [95% CI] |
| D 11 DV/I | XX/XX | [3/3/0/ 3/3/0/] |
| Durable PVI | (XX.X%) | [XX% - XX%] |
| I CDV about a included | XX/XX | [VV0/ VV0/] |
| LSPV chronic isolation | (XX.X%) | [XX% - XX%] |
| LIPV chronic isolation | XX/XX | [XX% - XX%] |
| LIF V CHIOIIC Isolation | (XX.X%) | |
| LCPV chronic isolation | XX/XX | [XX% - XX%] |
| LCF V chrome isolation | (XX.X%) | $\begin{bmatrix} \Lambda \Lambda / 0 - \Lambda \Lambda / 0 \end{bmatrix}$ |
| RSPV chronic isolation | XX/XX | [XX% - XX%] |
| KSF V chronic isolation | (XX.X%) | |
| RIPV chronic isolation | XX/XX | [XX% - XX%] |
| KIF V CHIOTIC ISOIATION | (XX.X%) | |
| RMPV chronic isolation | XX/XX | [XX% - XX%] |
| | (XX.X%) | $[\Lambda\Lambda/0 - \Lambda\Lambda/0]$ |
| CTI chronic isolation | XX/XX | [VV0/, VV0/,1 |
| C11 chronic isolation | (XX.X%) | [XX% - XX%] |
| LAPW chronic isolation | XX/XX | [XX% - XX%] |



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


# 4.1.6. Table 6. Per Remapped Veins Analysis

| | Veins Remapped $N = XX$ | |
|----------------------------------|-------------------------|-------------|
| | n/N (%) | [95% CI] |
| Number of veins durably isolated | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Number of veins with gaps | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Missing Data | XX | NA |

# 4.1.7. Table 7. Arrythmia Recurrence at 12 Months

| | ITT Population<br>N = XX | |
|---|---|---|
| | Mean±S.D. Median (min, max) (Q1, Q3) | [95% CI] |
| TTM compliance | XX±X<br>XX<br>(XX, XX)<br>(XX, XX) | [XX - XX] |
| | n/N (%) | [95% CI] |
| Holter compliance (6 month) | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Holter compliance (12 month) | | |
| Freedom from AF/AFL/AT | XX/XX<br>(XX.X%) | [XX% - XX%] |
| On AADs | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Off AADs | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Freedom from AF | XX/XX<br>(XX.X%) | [XX% - XX%] |
| On AADs | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Off AADs | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Freedom from AF/AFL/AT, no DCCV>90 days, no RF touch up, no ablation >90 days | XX/XX<br>(XX.X%) | [XX% - XX%] |
| On AADs | XX/XX | [XX% - XX%] |



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


| | (XX.X%) | |
|---|---|---|
| Off AADs | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Freedom from AF, no DCCV>90 days, no RF touch up, no ablation >90 days | XX/XX<br>(XX.X%) | [XX% - XX%] |
| On AADs | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Off AADs | XX/XX<br>(XX.X%) | [XX% - XX%] |

# 4.1.8. Table 8. Primary Safety Endpoint –Composite Safety Endpoint (CSE)

| | | opulation |
|--------------------------------------------------|---------|-----------|
| | | = XX |
| | n/N (%) | [95% CI] |
| Early and Late Onset Composite Safety Endpoint | XX/XX | [XX% - |
| | (XX.X%) | XX%] |
| Total Early (within 30 days of Index or Remap | XX/XX | [XX% - |
| Procedure) | (XX.X%) | XX%] |
| Death | XX/XX | [XX% - |
| | (XX.X%) | XX%] |
| Myocardial infarction (MI) | XX/XX | [XX% - |
| | (XX.X%) | XX%] |
| Persistent diaphragmatic paralysis | XX/XX | [XX% - |
| | (XX.X%) | XX%] |
| Stroke | XX/XX | [XX% - |
| | (XX.X%) | XX%] |
| Transient ischemic attack (TIA) | XX/XX | [XX% - |
| | (XX.X%) | XX%] |
| Peripheral or organ thromboembolism | XX/XX | [XX% - |
| - | (XX.X%) | XX%] |
| Pericarditis | XX/XX | [XX% - |
| | (XX.X%) | XX%] |
| Cardiac tamponade / perforation | XX/XX | [XX% - |
| | (XX.X%) | XX%] |
| Vascular access complications requiring | XX/XX | [XX% - |
| intervention | (XX.X%) | XX%] |
| Heart block | XX/XX | [XX% - |
| | (XX.X%) | XX%] |
| Total Late (any time during follow-up through 12 | XX/XX | [XX% - |
| months) | (XX.X%) | XX%] |
| Pulmonary vein (PV) stenosis (> 70% diameter | XX/XX | [XX% - |
| reduction from baseline) | (XX.X%) | XX%] |
| Atrio-esophageal fistula | XX/XX | [XX% - |
| | (XX.X%) | XX%] |



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


# 4.1.9. Table 9. Primary Feasibility Endpoint – Acute Procedural Success (ITT population)

| | ITT Population $N = XX$ | |
|---------------------------|-------------------------|-------------|
| | n/N (%) | [95% CI] |
| Acute Procedural Success* | XX/XX<br>(XX.X%) | [XX% - XX%] |

# 4.1.10. Table 10. Primary Feasibility Endpoint – Acute Procedural Success (PP population)

| | PP Population $N = XX$ | |
|---------------------------|------------------------|-------------|
| | n/N (%) [95% CI] | |
| Acute Procedural Success* | XX/XX (XX.X%) | [XX% - XX%] |

## 4.1.11. Table 11. Additional Endpoints

| | ITT Population $N = XX$ | |
|---|---|---|
| | Mean±S.D. Median (min, max) (Q1, Q3) | [95% CI] |
| Time to Therapeutic Failure (days) | XX±X<br>XX<br>(XX, XX)<br>(XX, XX) | [XX - XX] |
| | n/N (%) | [95% CI] |
| Proportion of subjects with Early recurrence of atrial fibrillation (ERAF) by 90 days after the index procedure | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Proportion of all ablated pulmonary veins that are isolated at the Index Procedure using the study device | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Proportion of all ablated pulmonary veins isolated using the study device during the Index Procedure that remain isolated at the 60-day remapping procedure | XX/XX<br>(XX.X%) | [XX% - XX%] |
| The proportion of attempted subjects that achieve Chronic CTI Success, defined as persistent bi-directional electrical block | XX/XX<br>(XX.X%) | [XX% - XX%] |



FARAPULSE\_PersAFOne II SAP V1.0 PERSAFONE II V1.0 Page 35 /42

| across the CTI assessed at the 60-day<br>Remapping Procedure | | |
|---|---|---|
| The proportion of attempted subjects that achieve Chronic Focal Success, defined as persistent electrical nonconductivity of all extra-PV tissue targeted for ablation in the Index Procedure, excluding the CTI, assessed at 60-day Remapping Procedure | XX/XX<br>(XX.X%) | [XX% - XX%] |

# 4.1.12. Table 12. Secondary Safety Endpoints

| | ITT Population $N = XX$ | |
|---|---|---|
| | n/N (%) | [95% CI] |
| Secondary Safety Endpoint (Early and Late<br>Onset Composite Safety Endpoint) assessed<br>at 7 days | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Total Early (within 7 days of Index or Remap Procedure) | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Death | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Myocardial infarction (MI) | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Persistent diaphragmatic paralysis | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Stroke | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Transient ischemic attack (TIA) | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Peripheral or organ thromboembolism | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Pericarditis | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Cardiac tamponade / perforation | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Vascular access complications requiring intervention | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Heart block | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Total Late (any time during follow-up through 12 months) | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Pulmonary vein (PV) stenosis (> 70% diameter reduction from baseline) | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Atrio-esophageal fistula | (XX/XX<br>(XX.X%) | [XX% - XX%] |



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


| Device-Related Serious Adverse Events (SAEs) | XX/XX<br>(XX.X%) | [XX% - XX%] |
|---|---|---|
| Procedure-Related Serious Adverse Events (SAEs) | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Stroke | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Transient Ischemic Attack (TIA) | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Cardioversion | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Arrhythmia-related (AF, AFL, AT) hospitalization | XX/XX<br>(XX.X%) | [XX% - XX%] |

# 4.1.13. Table 13. Secondary Feasibility Endpoints

| | ITT Population $N = XX$ | |
|---|---|---|
| | n/N (%) | [95% CI] |
| Chronic Procedural Success (CPS)* for subjects who undergo the protocolspecified 60-Day Remapping Procedure | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Acute Cavotricuspid isthmus (CTI) Success** | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Therapeutic Success*** | XX/XX<br>(XX.X%) | [XX% - XX%] |
| On AADs | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Off AADs | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Durability of the CTI and/or other extra PV lesion set(s) | | |
| Durability of CTI at remap | XX/XX<br>(XX.X%) | [XX% - XX%] |
| Durability of Mitral isthmus at remap | XX/XX<br>(XX.X%) | [XX% - XX%] |



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


| Durability of LAPW at remap | XX/XX<br>(XX.X%) | [XX% - XX%] |
|---|---|---|
| Durability of Left atrial roof line at remap | | |
| Durability of Left atrial Posterior line | | |

# 4.1.14. Table 14. Adverse Events (AEs) (not including SAEs)

| | $ ITT Population \\ N = XX $ | | |
|---|---|---|---|
| SOC Term/PT Term | Total<br>Number<br>of Events | Number of patients n | n/N (%)<br>[95% CI] |
| ALL | XX | XX | XX/XX |
| | | | (XX.X%) |
| | | | [XX% - |
| | | | XX%] |
| SOC1 | XX | XX | XX/XX |
| | | | (XX.X%) |
| | | | [XX% - |
| | | | XX%] |
| PT1 | XX | XX | XX/XX |
| | | | (XX.X%) |
| | | | [XX% - |
| | | | XX%] |
| PT2 | XX | XX | XX/XX |
| | | | (XX.X%) |
| | | | [XX% - |
| | | | XX%] |
| SOC2 | XX | XX | XX/XX |
| | | | (XX.X%) |
| | | | [XX% - |
| | | | XX%] |
| PT3 | XX | XX | XX/XX |
| | | | (XX.X%) |
| | | | [XX% - |
| 777.4 | 7777 | 7777 | XX%] |
| PT4 | XX | XX | XX/XX |
| | | | (XX.X%) |
| | | | [XX% - |
| | | | XX%] |



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


# 4.1.15. Table 15. Serious Adverse Events (SAEs)

| | ITT Population | | |
|---|---|---|---|
| | | N = XX | |
| SOC Term/PT Term | Total Number of Events | Number of patients n | n/N (%)<br>[95% CI] |
| ALL | XX | XX | XX/XX (XX.X%) [XX% -<br>XX%] |
| SOC1 | XX | XX | XX/XX (XX.X%) [XX% -<br>XX%] |
| PT1 | XX | XX | XX/XX (XX.X%) [XX% -<br>XX%] |
| PT2 | XX | XX | XX/XX (XX.X%) [XX% -<br>XX%] |
| SOC2 | XX | XX | XX/XX (XX.X%) [XX% -<br>XX%] |
| PT3 | XX | XX | XX/XX (XX.X%) [XX% -<br>XX%] |
| PT4 | XX | XX | XX/XX (XX.X%) [XX% -<br>XX%] |

## 4.1.16. Table 16. All Deaths

| | $\begin{array}{c} \text{ITT Population} \\ \text{N} = \text{XX} \end{array}$ | |
|---|---|---|
| | n/N (%) [95% CI] | |
| All-cause Mortality | XX/XX<br>(XX.X%) | [XX% - XX%] |

# 4.1.17. Table 17. Protocol Deviations according investigator without COVID-19

| | | ITT Population $N = XX$ | |
|---|---|---|---|
| Type of Deviation | Total Number of<br>Events | Number of patients n | n/N (%)<br>[95% CI] |
| Protocol Deviation Type 1 | XX | XX | XX/XX<br>(XX.X%)<br>[XX% - XX%] |
| Protocol Deviation Description 1 | XX | XX | XX/XX<br>(XX.X%)<br>[XX% - XX%] |
| Protocol Deviation Description n | XX | XX | XX/XX<br>(XX.X%) |



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


| | | | [XX% - XX%] |
|----------------------------------|----|----|-------------|
| | XX | XX | XX/XX |
| Protocol Deviation Type n | | | (XX.X%) |
| | | | [XX% - XX%] |
| | XX | XX | XX/XX |
| Protocol Deviation Description 1 | | | (XX.X%) |
| | | | [XX% - XX%] |
| | XX | XX | XX/XX |
| Protocol Deviation Description n | | | (XX.X%) |
| | | | [XX% - XX%] |

# 4.1.18. Table 18. Protocol Deviations according investigator with COVID-19

| | | ITT Population $N = XX$ | |
|---|---|---|---|
| Type of Deviation | Total Number of<br>Events | Number of patients n | n/N (%)<br>[95% CI] |
| Protocol Deviation Type 1 | XX | XX | XX/XX<br>(XX.X%)<br>[XX% - XX%] |
| Protocol Deviation Description 1 | XX | XX | XX/XX<br>(XX.X%)<br>[XX% - XX%] |
| Protocol Deviation Description n | XX | XX | XX/XX<br>(XX.X%)<br>[XX% - XX%] |
| Protocol Deviation Type n | XX | XX | XX/XX<br>(XX.X%)<br>[XX% - XX%] |
| Protocol Deviation Description 1 | XX | XX | XX/XX<br>(XX.X%)<br>[XX% - XX%] |
| Protocol Deviation Description n | XX | XX | XX/XX<br>(XX.X%)<br>[XX% - XX%] |

# 4.1.19. Table 19. Device Deficiency Summary Table

| | ITT Population<br>N = 25 |
|------------------------|----------------------------|
| Device deficiency rate | XX/XX (XX%)<br>[XX% - XX%] |



FARAPULSE\_PersAFOne II SAP V1.0 PERSAFONE II V1.0


# 4.2. Listings

4.2.17.

4.2.18.

| _ | |
|---|---|
| | isting 1: Patients populations, reasons of non-inclusion in the ifferent population, withdrawals and follow-up duration |
| 4.2.2. L | isting 2: Protocol deviations according the investigator |
| 4.2.3. L | isting 3: Demographics at baseline |
| 4.2.4. L | isting 4: AF History |
| 4.2.5. L | isting 5: Medical History (1/3) |
| 4.2.6. L | isting 6: Medical History (2/3) |
| 4.2.7. L | isting 7: Medical History (3/3) |
| 4.2.8. L | isting 8: Procedure data (1/4) |
| 4.2.9. L | isting 9: Procedure data (2/4) |
| 4.2.10. | Listing 10: Procedure data (3/4) |
| 4.2.11. | Listing 11: Procedure data (4/4) |
| 4.2.12. | Listing 12: Additional Ablation |
| 4.2.13. | Listing 13: Chronic Procedural Success at remap |
| 4.2.14. | Listing 14: Primary Safety endpoints |
| 4.2.15. | Listing 15: Device Deficiencies |
| 4.2.16. | Listing 16: Adverse events according CEC review |

Listing 17: Serious adverse events according CEC review

**Listing 18: Concomitant Medications** 



FARAPULSE\_PersAFOne II SAP V1.0 PERSAFONE II V1.0 Page 41 /42

# 4.3. Graphs

# 4.3.1. Graph 1: Patient disposition

# 4.3.2. Graph 2: Freedom from AF/AFL/AT on ADDs



## - Summary table

| | Group 1<br>(N=XXX) |
|---------------------------------|--------------------|
| Nb of patients | XXX |
| Nb of patients with an event | XX (XX.X%) |
| Nb of patients without an event | XX (XX.X%) |
| Survival rate | XX % |
| Time to event (days) | |
| Median | XX |
| (95% CI) | (XX, XX) |
| 25th-75th percentile | XXX – XXX |
| Range | X.XX - X.XX |



FARAPULSE\_PersAFOne II SAP V1.0

PERSAFONE II

V1.0


- 4.3.3. Graph 3: Freedom from AF/AFL/AT off ADDs
- 4.3.4. Graph 4: Freedom from AF on AADs
- 4.3.5. Graph 5: Freedom from AF off AADs
- 4.3.6. Graph 6: Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days
- 4.3.7. Graph 7: Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days on AADS
- 4.3.8. Graph 8: Freedom from AF/AFL/AT, no DCCV>90 days, no RF, no ablation >90 days off AADS
- 4.3.9. Graph 9: Freedom from AF, no DCCV>90 days, no RF, no ablation >90 days on AADs
- 4.3.10. Graph 10: Freedom from AF, no DCCV>90 days, no RF, no ablation >90 days off AADs
- 4.3.11. Graph 11: Death